CLINICAL TRIAL: NCT03528746
Title: The Acute Effect of Isometric Versus Isotonic Resistance Exercise in Patients With Patellar Tendinopathy: a Randomized, Participant Blinded, Crossover Trial
Brief Title: The Acute Effect of Isometric Versus Isotonic Resistance Exercise in Patients With Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Sinead Holden, Post- Doctoral Research Fellow, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: N-20160084
Record Dates: First submitted 2017-12-05; First posted 2018-05-18 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Patellar Tendinitis
Keywords: Patellar tendinopathy
MeSH Terms: interventions — Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: The proposed study is a participant blinded, randomised crossover superiority trial, to examine acute effect of isometric versus isotonic resistance exercise on pain in patients with patellar tendinopathy.
Who Masked: Participant
Masking Description: Participants will be blinded to the study hypothesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercise (Experimental): Participants will complete isometric quadriceps exercise
  Interventions: Other: Isometric exercise
- Isotonic exercise (Active Comparator): Participants will complete dynamic leg extension
  Interventions: Other: Isotonic Exercise

INTERVENTIONS:
Other: Isotonic Exercise — Participants will complete dynamic leg extension in a leg extension machine with a range of motion from approximately 90 degrees flexion to full extension. Each repetition will be completed with a 3s concentric contraction, 0s isometric and 4s eccentric contraction.This will be repeated for 8 repetitions and for 5 sets with 2 minutes rest between each set, as per Rio and colleagues. The load used during the isotonic exercise will be equivalent to participants 8 repetition maximum, which will be determined by an experienced tester in a standardised manner according to NSCA guidelines.
  Other Names: resistance exercise
  Arms: Isotonic exercise
Other: Isometric exercise — Participants will complete isometric quadriceps exercise, where they must hold a load statically for 45s with their knee in 60° flexion. This will be repeated for 5 sets with 2 minutes rest between each set. A load of 70% of the maximal voluntary isometric contraction (MVIC) will be used. MVIC will be assessed in an isokinetic dynamometer as per Rio and colleagues. Participants will be seated in a stable position in the dynamometer with the knee at 60° of knee flexion. First they will be familiarised with the procedure. Standardised instructions will be issued for participants to perform a maximal effort knee extension against the dynamometer for 3seconds. After a short break, the test will be repeated three times and the MVIC will be peak torque recorded during these three efforts.
  Arms: Isometric exercise

SUMMARY:
The purpose of this study is to compare the acute effects of two different types of resistance exercise (isometric versus isotonic) on exercise induced hypoalgesia during an aggravating activity, in participants with patellar tendinopathy.

DETAILED DESCRIPTION:
Exercise is a commonly prescribed treatment for patients with musculoskeletal pain, and is effective in treating tendon pain. It is well documented, that an acute bout of aerobic or resistance type exercise reduces sensitivity to pain in healthy individuals. Therefore the efficacy of exercise as an intervention may be partially due to the analgesic effect of exercise, also termed exercise-induced hypoalgesia (EIH).

For tendinopathies, high load resistance exercise is frequently used during rehabilitation.

However, the optimal mode and dosages required for reducing pain in patients with tendinopathies is unknown. Understanding the effect of different forms of exercise on pain may help optimize the prescription of exercise for pain management.

A recent study by Rio and colleagues documented the acute effect of two different forms of resistance exercise in patients with patellar tendinopathy. The study compared, isometric resistance exercise (static muscular contractions), in comparison to isotonic resistance exercise (dynamic contractions) and found that isometric exercise induced greater participantive pain relief in response to an aggravating task. This study was the first to compare the analgesic effect of different forms of resistance exercise in patients with tendinopathy.

Although the results appear promising, a limitation of the study was that it did not quantify the effect of the different exercises on measures of pain sensitivity as in previous studies examining EIH.

Purpose The purpose of this study is to compare the acute effects of two different types of resistance exercise (isometric versus isotonic) on exercise induced hypoalgesia during an aggravating activity, in participants with patellar tendinopathy.

Hypothesis The primary hypothesis is that isometric exercise will induce greater pain relief/reduction during an aggravating activity in comparison to isotonic exercises.

Study Design and Methods The proposed study is a participant blinded, randomised crossover superiority trial, to examine acute effect of isometric versus isotonic resistance exercise on pain in patients with patellar tendinopathy. The trial will be pre-registered on clinicaltrials.gov before inclusion of participants commences.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-40 years, with patellar tendinopathy will be included. Diagnosis of patellar tendinopathy, will be made by a physiotherapist (who has been trained by an experienced rheumatologist) as follows, similar to previously outlined criteria:

  * pain localised to the inferior pole of the patella during jumping and landing activities
  * pain during testing on the single-leg decline squat (SLDS)
  * The diagnosis will be confirmed by the presence of characteristic features on ultrasound imaging (eg, hypoechoic area and focal enlarged tendon).
  * Minimum pain of 3cm on a 10cm visual analogue scale (VAS)
  * Other concurrent diagnosable knee pathologies

Exclusion Criteria:

* Previous surgery of the knee
* Pregnancy
* Corticosteroid injection within the previous 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Change in pain during aggravating activity | baseline; immedietely after exercise
  The single leg decline squat (SLDS) will be used as the provocative activity, as this is an activity that usually induces pain in patients with patellar tendinopathy. Participants will be asked to stand on one limb, with their heel raised, so they are in approximately 25 degrees of plantar flexion. They will then be asked to perform a small squat, to about 60 degrees of knee flexion. This will be repeated three times. Participants will provide a numerical pain rating score for the decline squat on an 11-point numerical rating scale (NRS), anchored at left with '0, no pain' and at right with '10, worst possible pain'. If participants have bilateral patellar tendinopathy, data from the 'most painful' limb (indicated by participants) will be used for the primary outcome.

SECONDARY OUTCOMES:
change in pain during aggravating activity | baseline; 45 minutes post exercise
  The single leg decline squat (SLDS) will be conducted as above.
change in pressure pain threshold (kPa) | Baseline; Immediately after exercise; 45 min post exercise
  Pain sensitivity is examined by the participants' pressure pain threshold (PPT). A hand-held algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe (covered by a disposable latex sheath) will be used to record the PPT. The probe is placed perpendicular to the skin and pressure is increased gradually at a rate of 30 kPa/s. Participants will be instructed to indicate when the sensation first changes from a sensation of pressure, to a sensation of pressure pain. The patient is fitted with a hand-held switch and is instructed to press the switch as soon as the pressure triggers pain, stopping the pressure algometer. To determine local pain sensitivity, PPTs will be done, at the most painful site point on the tendon as per previously methods in patellar tendionopathy which have demonstrated reliability. PPTs will also be taken at a distal site (on the muscle of tibialis anterior) to reflect segmental hypoalgesia and remotely at the elbow.
Change in patellar tendon thickness (mm) | Baseline; Immedietly after exercise
  Patellar tendon thickness will be measured by ultrasonography

OTHER OUTCOMES:
Pain (during exercise) | Immediately after exercise set
  Participants will provide a numerical pain rating score on an 11-point numerical rating scale (NRS), anchored at left with '0, no pain' and at right with '10, worst possible pain'.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available from the PI upon reasonable request.

REFERENCES:
- [Background] Rio E, Kidgell D, Purdam C, Gaida J, Moseley GL, Pearce AJ, Cook J. Isometric exercise induces analgesia and reduces inhibition in patellar tendinopathy. Br J Sports Med. 2015 Oct;49(19):1277-83. doi: 10.1136/bjsports-2014-094386. Epub 2015 May 15. PMID 25979840